CLINICAL TRIAL: NCT00413504
Title: Fondaparinux as Monotherapy for Deep Vein Thrombosis and/or Pulmonary Embolism (Pilot Study)
Brief Title: Fondaparinux as Monotherapy for DVT and/or Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Brigham and Women's Hospital, Venous Thromboembolism Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000599
Record Dates: First submitted 2006-12-07; First posted 2006-12-19 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Fondaparinux; Monotherapy; Deep Vein thrombosis; Pulmonary Embolism; Anticoagulation
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fondaparinux

SUMMARY:
To determine whether fondaparinux as monotherapy without warfarin is effective and safe for long-term (90 days) treatment of DVT and/or PE, thus gaining new long-term experience and data using fondaparinux.

DETAILED DESCRIPTION:
Background and Significance:

Warfarin is usually prescribed to manage long-term anticoagulation of deep vein thrombosis (DVT) and pulmonary embolism (PE). However about 5% of patients are unable to tolerate warfarin or to be safely or effectively anticoagulated. Some of the reasons for discontinuing warfarin anticoagulation and switching patients to parenteral anticoagulation are as follows:

1. Recurrent venous thromboembolism despite anticoagulation with warfarin
2. Clinically important bleeding complications due to warfarin
3. Inability to achieve target International Normalized Ratio (INR) on warfarin
4. Nonbleeding side effects of warfarin, such as hair loss or rash.

These patients who cannot tolerate or respond adequately to warfarin are usually managed with "off-label" twice-daily enoxaparin injections as monotherapy. The approved duration of treatment of DVT and PE with fondaparinux is 5 to 9 days as a "bridge" to warfarin. Until now, no studies have investigated the use of fondaparinux for more than 26 days for the treatment of PE and more than 10 days for the treatment of DVT.

Treatment doses of twice-daily enoxaparin are only Food and Drug Administration (FDA) approved for 5 to 14 days for "bridging" for the treatment of acute DVT and/or PE patients to warfarin.

Fondaparinux is a synthetic antithrombotic agent with specific anti-factor Xa activity. Its pharmacokinetic properties allow for a simple, fixed-dose, once daily regimen of subcutaneous injection, without the need for dose adjustment based on laboratory monitoring.

Fondaparinux is available only in 3 treatment doses and is prescribed once every 24 hours based on patient's weight: 5 mg for patients weighing less than 50 kg, 7.5 mg for patients weighing between 50 to 100 kg, and 10 mg for patients weighing more than 100 kg and is available in prefilled syringes. Also, fondaparinux does not cross react with heparin-induced platelet antibodies, and heparin-induced thrombocytopenia has never been documented with fondaparinux.

The MATISSE Investigators showed that once-daily, subcutaneous administration of fondaparinux for at least 5 days and until 2 consecutive INRs were greater than 2.0 as a "bridge" to warfarin is at least as effective and safe as adjusted-dose, intravenous administration of unfractionated heparin as a "bridge" to warfarin in the initial treatment of hemodynamically stable patients with pulmonary embolism. During the 3-month follow up, 42 of the 1103 patients randomly assigned to receive fondaparinux (3.8 percent) had recurrent thromboembolic events, as compared with 56 of the 1110 patients randomly assigned to receive unfractionated heparin (5.0 percent). Major bleeding occurred in 1.3 percent of the patients treated with fondaparinux and 1.1 percent of those treated with unfractionated heparin. Mortality rates at three months were similar in the two groups.

In another randomized double-blinded trial by the MATISSE Investigators, patients were randomized to fondaparinux once daily versus enoxaparin twice daily for at least 5 days and until 2 consecutive INRs were greater than 2.0 as a "bridge" to warfarin for initial treatment of acute symptomatic DVT. Fondaparinux was found to be as effective and safe as twice-daily enoxaparin during the 3-month follow up period. 43 (3.9%) of 1098 patients randomly assigned to fondaparinux had recurrent thromboembolic events compared with 45 (4.1%) of 1107 patients randomly assigned to enoxaparin. Major bleeding occurred in 1.1% of patients receiving fondaparinux and 1.2% of patients receiving enoxaparin. Mortality rates were 3.8% and 3.0%, respectively.

These two MATISSE trial totaled 4418 patients and led to the FDA approval of fondaparinux in the treatment of acute symptomatic DVT and PE as a "bridge" to warfarin.

In this investigator-initiated trial, we will conduct a cohort study with once daily fondaparinux as monotherapy without warfarin for 90-day management of DVT and/or PE in patients who are unable to tolerate or respond adequately to warfarin.

Research Design and Methods:

This is a cohort study with a sample size of 30 patients at Brigham and Women's Hospital with history of DVT and/or PE who are intolerant to warfarin or not responding to warfarin.

During the study there will be 3 visits at day zero, week 6, and at day 90. Patients will be monitored closely for any bleeding complications.

During these visits, blood will be drawn for platelet counts, renal function, hematocrit, and transaminase level.

Primary endpoints

1. Recurrent acute symptomatic DVT confirmed by venous ultrasound and/or CT scan
2. Recurrent acute symptomatic PE confirmed by chest CT scan
3. Major hemorrhage defined as spinal, retroperitoneal or intracranial bleeding, drop in hemoglobin ≥2g/dl or transfusion ≥2U or surgical or medical intervention, death related to bleeding

Secondary endpoints

Comparison of Day Zero, 6 week, and Day 90 platelet counts, renal function, hematocrit and transaminase level

Drug Dose:

Patients enrolled in the study will receive a weight-based dose of fondaparinux as monotherapy for 90 days for the treatment of DVT and/or PE.

Weight < 50 kg - 5 mg daily Weight 50 - 100 kg - 7.5 mg daily Weight > 100 kg - 10 mg daily

Biostatistical Analysis:

Descriptive statistics will be performed using age, gender, and indication for long-term anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent venous thromboembolism despite anticoagulation with warfarin(Or)
2. Clinically important bleeding complications due to warfarin(Or)
3. Inability to achieve the target INR on warfarin(Or)
4. Nonbleeding side effects of warfarin, such as hair loss, rash, purple toe syndrome(Or)
5. Patient with cancer on monotherapy with parenteral anticoagulation for DVT and/ or PE

   and
6. Require at least 90 days of anticoagulation
7. Require anticoagulation for objectively confirmed DVT and/or PE
8. Age greater than 18 years
9. Written informed consent

Exclusion Criteria:

1. Patients with renal insufficiency, defined as creatinine > 1.5 mg/dl
2. Patients in whom anticoagulation with any agent is deemed unsafe due to bleeding risk.
3. Pregnancy
4. Known hypersensitivity to fondaparinux

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Recurrent acute symptomatic DVT confirmed by venous ultrasound and/or CT scan | 90 Days
Recurrent acute symptomatic PE confirmed by chest CT scan | 90 Days
Major hemorrhage defined as spinal, retroperitoneal or intracranial bleeding, drop in hemoglobin ≥2g/dl or transfusion ≥2U or surgical or medical intervention, death related to bleeding | 90 Days

SECONDARY OUTCOMES:
Comparison of Day Zero, 6 week, and Day 90 platelet counts, renal function, hematocrit and transaminase level | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Petitou M, Duchaussoy P, Herbert JM, Duc G, El Hajji M, Branellec JF, Donat F, Necciari J, Cariou R, Bouthier J, Garrigou E. The synthetic pentasaccharide fondaparinux: first in the class of antithrombotic agents that selectively inhibit coagulation factor Xa. Semin Thromb Hemost. 2002 Aug;28(4):393-402. doi: 10.1055/s-2002-34309. PMID 12244487
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, van den Berg-Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Subcutaneous fondaparinux versus intravenous unfractionated heparin in the initial treatment of pulmonary embolism. N Engl J Med. 2003 Oct 30;349(18):1695-702. doi: 10.1056/NEJMoa035451. PMID 14585937
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Fondaparinux or enoxaparin for the initial treatment of symptomatic deep venous thrombosis: a randomized trial. Ann Intern Med. 2004 Jun 1;140(11):867-73. doi: 10.7326/0003-4819-140-11-200406010-00007. PMID 15172900
- See also: North American Thrombosis Forum — http://www.natfonline.org